CLINICAL TRIAL: NCT06756919
Title: EFFECTS OF MUSIC THERAPY DURING ENDOSCOPY ON PAIN, ANXIETY AND VITAL SIGNS: A RANDOMIZED CONTROLLED STUDY
Brief Title: EFFECTS OF MUSIC THERAPY DURING ENDOSCOPY ON PAIN, ANXIETY AND VITAL SIGNS
Acronym: MUSCOPY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Şerife Naz Bozkurt, Principal Investigator, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2023/176
Record Dates: First submitted 2024-12-24; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Music Therapy
Keywords: music; endoscopy; nursing; pain; vital signs
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients Having Endoscopy with Music Therapy (Experimental): Patients having endoscopy procedure with music therapy
  Interventions: Behavioral: Music intervention
- Control Group (No Intervention): Patients having endoscopy without music therapy

INTERVENTIONS:
Behavioral: Music intervention — Music therapy ( nature sounds) during the endoscopy procedure
  Arms: Patients Having Endoscopy with Music Therapy

SUMMARY:
This study was conducted to evaluate the effect of music therapy on the vital signs, anxiety and pain of the patients during endoscopy procedure

DETAILED DESCRIPTION:
The aim of this study was to the effects of music during the endoscopy procedure on anxiety, pain and vital signs.This study was conducted as a randomized, controlled, double-blind trial. The study population consisted of patients in the endoscopy unit of a university hospital between June and December 2023. The patients were randomly divided into the experimental group, who listened to music during endoscopy, and the control group, which did not receive any intervention other than routine nursing care. This study, data were collected via a patient information form, the State-Trait Anxiety Inventory (STAI-State), the visual analogue scale (VAS), and a vital signs monitoring form.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have endoscopy procedure
* Being older than 18 years old
* Not having hearing problems
* ASA status between 1-3

Exclusion Criteria:

* Cognitive or psycological disorders
* Regular usage of analgesic/anxiolytic/sedaditive drugs
* Haemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
State-trait anxiety inventory | 6 months
Visual Analog Scale | 6 months
Patient Information Form | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No